CLINICAL TRIAL: NCT02007148
Title: MetronomIc CApecitabine and DOcetaxel as Second-line Chemotherapy for Advanced Gastric Cancer Patients Previously Treated With Fluoropyrimidine and Platinum Agents MiCADO Study
Brief Title: MetronomIc CApecitabine and DOcetaxel as Second-line Chemotherapy for Advanced Gastric Cancer
Acronym: MICADO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Group of Endovascular Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MICADO01; MICADO (Other: IGEVO)
Record Dates: First submitted 2013-11-29; First posted 2013-12-10 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: gastric adenocarcinoma,; capecitabine,; second line treatment,; recurrent or metastatic disease,; overall survival,; tumor response,; quality of life
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- micado (Experimental): CAPECITABINE 500 mg twice a day, orally, continuously DOCETAXEL 60 mg/sqm i.v. over 1 hr on day 1 cycles repeated every 3 weeks Duration of treatment: Chemotherapy should be continued until: progressive disease; unacceptable toxicities; patients' refusal; or upon investigator's judgement is in the best interest for the patient.
  Interventions: Drug: capecitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: capecitabine — twice a day
  Other Names: xeloda
Drug: Docetaxel — cycles repeated every 3 weeks
  Other Names: taxotere

SUMMARY:
Second-line chemotherapy represents an option in gastric cancer, especially for patients with adequate performance status. Two randomized phase III trials comparing 2nd-line docetaxel with best-supportive care have reported a benefit in favor of chemotherapy. Capecitabine is a fluoropyrimidine carbamate, which has a broader spectrum of antitumor activity than other fluoropyrimidines. In gastric cancer xenografts. metronomic capecitabine inhibited angiogenesis, growth of gastric cancer and improved survival with less toxicity. Given its potential low toxicity, the combination of docetaxel and metronomic capecitabine needs to be evaluated to assess efficacy and tolerability in patients with advanced gastric cancer previously treated with a fluoropyrimidine-based and platinum-based chemotherapy.

DETAILED DESCRIPTION:
Despite a declining incidence in many developed countries, gastric cancer remains the second most common cause of cancer deaths, and it is responsible for about 12% of all cancer-related deaths worldwide. More than two-thirds of patients diagnosed with gastric cancer will have unresectable disease and despite the fact that surgical pathological resection can be curative for many patients, most of them develop recurrent disease. Evidence supports the use of palliative chemotherapy with the aims of improving symptoms, quality of life, and possibly prolonging survival. Combination chemotherapy regimens have been developed in the hopes of improving response rate and overall survival (OS). Unfortunately, the benefits of combination chemotherapy have been modest. In general, regimens containing fluoropyrimidine and platinum agents are widely accepted as potential standard therapies. Although a large proportion of patients with metastatic or recurrent gastric cancer may initially respond to chemotherapy, they ultimately progress. In addition, many patients have primary refractory disease. The median survival at progression after first-line chemotherapy for metastatic gastric cancer is about 2.5 months.

Docetaxel is one of the most active single agents in the treatment of gastric cancer. In the first line setting, at a dose of 60-100 mg/m2 repeated every 3 weeks, response rates ranged from 17% to 20%. Docetaxel is the only taxane that has been evaluated in the context of a phase III study.

Low-dose metronomic chemotherapy represents a new strategy to treat solid tumors by exhibiting stronger anti-angiogenic activity and less side effects, especially in combination with other anti-angiogenic agents. Capecitabine is a fluoropyrimidine carbamate, which has a broader spectrum of antitumor activity than other fluoropyrimidines. In gastric cancer xenografts. metronomic capecitabine inhibited angiogenesis, growth of gastric cancer and improved survival with less toxicity. In combination with other drugs, the treatment with metronomic capecitabine has proven its efficacy with minimal toxicity in breast cancer, in metastatic renal-cell carcinoma, in advanced adrenocortical carcinoma, in hepatocellular carcinoma, in prostate cancer.

The "metronomic" strategy was also considered in pretreated elderly patients with advanced gastric cancer. Eligible patients with advanced gastric cancer were treated with capecitabine until disease progression or significant toxicity. Metronomic chemotherapy achieved a disease control rate at 8 weeks of 51.1% , and the objective response rate was 20.9% . The median time-to-progression and median overall survival were 3.6 months and 7.6 months, respectively. Grade II neutropenia and thrombocytopenia were observed in 13.3 and 2.2% of patients, respectively. Grade II/III nonhematological toxicities included diarrhea (4.4%), stomatitis (13.4%), and hand-foot syndrome (15.5%). No grade 4 toxicity, neutropenic fever or treatment-related deaths occurred.

Based on these premises and to the fact that the role of metronomic chemotherapy remains controversial, its optimal therapeutic use has not yet been defined, we designed this phase II study with tha aim to assess efficacy and tolerability of metronomic capecitabine in combination with the conventional use of docetaxel in patients with advanced gastric cancer previously treated with a fluoropyrimidine-based and platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Histologically or cytologically confirmed gastric adenocarcinoma, including gastric or gastroesophageal-junction adenocarcinoma (GEJ)
3. Measurable disease based on computed tomography
4. Eastern Cooperative Oncology Group performance status 0 or 1
5. Treatment with only 1 prior regimen (as first-line therapy) that must have included a fluoropyrimidine and a platinum agent
6. Disease progression after the start of the prior regimen based on computed tomography (or magnetic resonance imaging in the event of allergy to contrast medium)
7. Adequate bone marrow, hepatic, and renal function,
8. At least 4 weeks and recovery from effects of prior major surgery or radiation therapy
9. If previously administered as treatment for gastric cancer, prior to study entry a washout period equivalent to at least 5 half-lives for antibodies and of at least 28 days for chemotherapy (Concurrent use of bisphosphonates is permitted.)
10. Ability to swallow an oral solid-dosage form of medication, including when a feeding tube is present
11. A negative serum pregnancy test within 7 days prior to accrual in women of childbearing potential
12. Agreement to use an effective form of contraception
13. Signed written informed consent.
14. Ability to comprehend and to comply with the requirements of the study.

Exclusion Criteria:

1. Squamous cell gastric carcinoma
2. Bone-only metastatic disease
3. History or presence of brain metastasis or leptomeningeal disease
4. Operable gastric or GEJ cancer
5. Herceptin 2 (HER2) -positive disease if the subject has not previously been treated with an anti-HER2 agent
6. Uncontrolled diarrhea, defined as more than 3 loose bowel movements above the subject's usual number of bowel movements on at least 3 days within the 14 days prior to study entry
7. Nausea or vomiting for at least 3 consecutive days within the 14 days prior to study entry despite the administration of standard antiemetic therapy
8. Known malabsorptive disorder
9. Second cancer (except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the subject has been disease-free for 5 or more years)
10. Human immunodeficiency virus infection based on history of positive serology
11. Significant medical disease other than gastric cancer, including but not limited to uncontrolled diabetes mellitus, active angina or heart failure, uncontrolled hypertension, or an active psychiatric condition that would prevent consistent and compliant participation in the study
12. Presence of neuropathy > Grade 1
13. Prior treatment including docetaxel
14. Prior radiation therapy to more than 25% of the bone marrow
15. Need for other anticancer treatment (such as chemotherapy, radiation therapy, or biologic therapy with an approved or investigational agent) while receiving protocol therapy
16. History of severe or unexpected reaction to fluoropyrimidine therapy
17. History of hypersensitivity to fluoropyrimidine agents or any of their ingredients.
18. Known dihydropyrimidine dehydrogenase deficiency
19. Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2013-11; Primary Completion 2021-10 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
tumor response | 6 months
  CT scan evaluated with RECIST 1.1

SECONDARY OUTCOMES:
progression-free survival | 6 months
  progression-free survival
overall survival | 12 months
  overall survival
number of patients with Adverse Events | 6 months
  number of patients with Adverse Events
time to treatment failure | 6 months
  time to treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Catalano, MD, Principal Investigator — AORMN, U.O.C. Oncologia, Ospedale San Salvatore
Locations (2):
- Italy (2):
  - AORMN, Presidio Ospedaliero San Salvatore, Pesaro
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio Ospedaliero San Salvatore, Pesaro

REFERENCES:
- [Background] Cascinu S, Graziano F, Barni S, Labianca R, Comella G, Casaretti R, Frontini L, Catalano V, Baldelli AM, Catalano G. A phase II study of sequential chemotherapy with docetaxel after the weekly PELF regimen in advanced gastric cancer. A report from the Italian group for the study of digestive tract cancer. Br J Cancer. 2001 Feb;84(4):470-4. doi: 10.1054/bjoc.2000.1631. PMID 11207039
- [Background] Graziano F, Catalano V, Baldelli AM, Giordani P, Testa E, Lai V, Catalano G, Battelli N, Cascinu S. A phase II study of weekly docetaxel as salvage chemotherapy for advanced gastric cancer. Ann Oncol. 2000 Oct;11(10):1263-6. doi: 10.1023/a:1008373814453. PMID 11106114
- [Background] Catalano V, Labianca R, Beretta GD, Gatta G, de Braud F, Van Cutsem E. Gastric cancer. Crit Rev Oncol Hematol. 2009 Aug;71(2):127-64. doi: 10.1016/j.critrevonc.2009.01.004. Epub 2009 Feb 20. PMID 19230702
- [Background] Catalano V, Vincenzi B, Giordani P, Graziano F, Santini D, Baldelli AM, Alessandroni P, Schiavon G, Rossi D, Casadei V, D'Emidio S, Luzi Fedeli S, Tonini G, Fiorentini G. Sequential chemotherapy with cisplatin, leucovorin, and 5-fluorouracil followed by docetaxel in previously untreated patients with metastatic gastric cancer: a phase II study. Gastric Cancer. 2012 Oct;15(4):419-26. doi: 10.1007/s10120-011-0134-1. Epub 2012 Jan 12. PMID 22237659
- See also: International group of endovascular oncology (IGEVO) website — http://igevo.jimdo.com/